CLINICAL TRIAL: NCT01758536
Title: A Phase IV, Double Blind, Placebo-controlled, Randomized, Multi-Center Study to Evaluate the Efficacy of Huatuo Zaizao Pills in Improving of Neural Function in Acute Ischemic Stroke
Brief Title: Efficacy Study of Huatuo Zaizao Pills in Improving of Neural Function in Acute Ischemic Stroke
Acronym: HTZZP-INF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Guangzhou Baiyunshan Qixing Pharmarceutical Co Ltd (Unknown)
Responsible Party: Principal Investigator, Qiang Dong, Professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QIXING-2012
Record Dates: First submitted 2012-12-24; First posted 2013-01-01 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; neural function; life quality
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Pills (Placebo Comparator): * 12 g each time, twice daily.
  * 3 months
  Interventions: Drug: Huatuo Zaizao Pills
- Huatuo Zaizao Pills (Experimental): * 12 g each time, twice daily.
  * 3 months.
  Interventions: Drug: Huatuo Zaizao Pills

INTERVENTIONS:
Drug: Huatuo Zaizao Pills — A tens of herbs botanical drug product 12 gram (g) in 72 mini pills formulation. It is to be used as 12 g each time, twice daily.
  Other Names: Huatuo Zaizao Wan

SUMMARY:
The purpose of this study is to determine the efficacy of Huatuo Zaizao Pills in improving neural function and life quality in patients with acute ischemic stroke in China.

DETAILED DESCRIPTION:
Huatuo Zaizao Pills is a pure natural preparation from plant origin and consists of Chuanxiong rhizome, Evodia fruit and etc. Most of its ingredients are not opened and reserved by the National Commission for Science and Technology and the State Food and Drug Administration.

Huatuo Zaizao Pills was approved for marketing as a drug over several decades for treating and preventing cardiovascular and cerebrovascular diseases and their sequela. It is used to symptoms induced by blood stasis or stagnation of phlegm-wetness, such as stroke and paralysis, stiffness and numbness, deviation of the eye and mouth and dysphasia.

Based on the history of Huatuo Zaizao Pills for the treatment of cerebral infarction and hemorrhagic stroke, investigators will perform a phase IV, double blind, placebo-controlled, randomized and multi-Center clinical trial in China to determine the efficacy of Huatuo Zaizao Pills in improving neural function and life quality in patients with acute ischemic stroke in China.

The study was designed with a target sample size of 1100 patients and the investigators will perform 200 patients in the first period. Patients will be randomly assigned to receive Huatuo Zaizao Pills or placebo at dose of 12g each time, twice daily.

The investigators hypothesis that this study might offer based medicine evidence to test and verified the efficacy of Huatuo Zaizao Pills in improving the neural function and life quality in patients with ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be between the ages of 18 and 70 years.
* Patient must be with ischemic stroke and at stroke onset 14th day.
* Patient must be with mRS score <5 at enrollment and mRS score ≤1 before stroke onset.
* Symptoms and imaging of CT (computed tomography) or MRI (Magnetic Resonance Imaging) support the diagnosis of ischemic stroke.
* Patient must be with 4 ≤ NIHSS ≤16.
* Patient must be with Glasgow coma scale (GCS) ≥7.
* Only patient with an anterior circulation infarction of Oxfordshire Community Stroke Project (OCSP)classification and atherothrombosis or cardioembolism of modified TOAST classification were accepted.
* Patient must understand and be willing, able and likely to comply with all study requirements.
* Informed consent must be obtained.

Exclusion Criteria:

* Patient with severe cognitive impairment who not be able to give voluntary written informed consent or participate in this study.
* Maybe not to comply with all study requirements or not be able to participate in this study for regional or social reasons.
* Pregnancy, breast feeding and the possible pregnancy during study.
* Participating in another medicine or interference study in the same time or at least within 3 months, or enrolled in this study in other location.
* Patient with mRS≥5 at enrollment.
* Coma patient with GCS<7.
* Patient with severe cerebral function impairment which was not caused by stroke.
* Patient with dysphagia, Wyatt score ≥2.
* Lacunar infarction.
* Patient accompanied with systemic diseases: gastrointestinal hemorrhage, advanced carcinoma, liver malfunction, kidney malfunction, severe dementia or mental disorder.
* Unstable patient after receiving thrombolytic therapy.
* Cerebral hemorrhage verified by CT or MRI.
* History of major operation or trauma within 6 weeks or having a major operation arrangement.
* Allergic to one or more components of study medicine.
* Receiving study medicine or components of study medicine within 2 weeks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale | 3 months
  The primary end point is the proportion of patients with a modified Rankin Scale (mRS) score of 0 to 1 at 3 months.

SECONDARY OUTCOMES:
modified Rankin Scale,NIHSS, Barthel Index, and MMSE | 3 months
  * The proportion of patients with a modified Rankin Scale (mRS) score of 0 to 2 at 3 months.
  * NIHSS (National Institute of Health Stroke Scale) score.
  * The proportion of patients with BI no less than 75 at 3 months.
  * MMSE(Mini-Mental State Examination)score.

OTHER OUTCOMES:
Traditional Chinese Symptoms and tongue image | the first day of enrollment
  Recording the Traditional Chinese Symptoms and taking tongue photo for traditional Chinese doctors to perform subgroup analysis

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Dong, MD, Principal Investigator — Huashan Hospital
Locations (4):
- China (4):
  - Huashan Hospital, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - Shanghai Shuguang Hospital, Shanghai